CLINICAL TRIAL: NCT06067360
Title: Hydrodissection Sleeve to Aid Cataract Surgery
Brief Title: Evaluation of Performance of New IFIS Sleeve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medicel AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFIS2023
Record Dates: First submitted 2023-09-21; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sleeve (Experimental): Evaluation of IFIS sleeve performance
  Interventions: Device: IFIS sleeve

INTERVENTIONS:
Device: IFIS sleeve — IFIS sleeve will be inserted to prevent iris prolapse

SUMMARY:
A silicone sleeve will be used on the hydrodissection needle to avoid that the iris can prolaps through the gap between needle and incision wound.

DETAILED DESCRIPTION:
Cataract surgey is a common operation approximately 25 million pocedures per year worldwide. An essential step of the procedure is hydrodissection where fluid is forced into the eye through a cannula to free the cataract from its capsule. A serious and potential sight threatening complication of hydrodissection is iris prolapse, where the iris comes out of the wound. The overall incidence of iris prolapse during cataract surgery is 0.9% and higher in patients with intraoperative floppy iris syndrome (IFIS) at 11.9% , small pupils and small eyes. Patients on Tamsulosin medication with a Full Set of Project Data IRAS Version 6.3.3 5 DRAFT pupil less than 7.5mm have a 79% risk of prolapse Iris prolapse most often occurs during hydrodissection because the hydrodissection cannula is smaller (approx.1mm) than the wound (2.2-2.7mm) it is introduced through. Therefore the iris can be forced out / prolapse through this gap by the forced injection of fluid.

Traditional methods such as phenylephrine injection into the eye have varying effects can be unlicensed and possibly increase the prolapse risk. Mechanical pupil stretching can permanently damage the iris with complications.

Phacosleeve hydrodissection where the wound is sealed by a phacosleeve and the hydrodissecting irrigation cannula introduced through the sleeve or from side port /incison. The phacosleeve is not designed for this. This study is to use a purpose made tapered sleeve by Medicel in the same fashion as the current phacosleeve.

ELIGIBILITY:
Inclusion Criteria:

* patient with planned cataract surgery

Exclusion Criteria:

* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
performance of IFIS sleeve to prevent iris prolapse | The evaluation of the device is during cataract surgery, which typically is less than 10 minutes. No additional treatments or evaluations after the surgery.
  performance of the IFIS sleeve to successfully prevent from iris prolapse: Iris prolaps is a distinct complication that can occurr during cataract surgery. For each treatment, the surgeon will protocol, whether a prolaps occurred during the surgical procedure. The primary outcome is the number of prolaps cases over all surgeries.

IPD SHARING:
Plan to Share IPD: No